CLINICAL TRIAL: NCT02887807
Title: CYclosporine A in Shockable Out-of-hospital Cardiac Arrest ResUScitation
Acronym: CYRUS II
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-753
Record Dates: First submitted 2016-08-18; First posted 2016-09-02 (Estimated); Last update posted 2019-03-14 (Actual); Status verified 2019-03

CONDITIONS: Shockable Out of Hospital Cardiac Arrest
Keywords: Cardiac arrest; Shockable; Cyclosporine
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cyclosporine A (Experimental): Single intravenous bolus of cyclosporine A (2.5 mg/kg) at the onset of resuscitation
  Interventions: Drug: Single intravenous bolus of cyclosporine A (2.5 mg/kg) at the onset of resuscitation
- Control (Placebo Comparator): Single intravenous bolus of placebo (2.5 mg/kg) at the onset of resuscitation
  Interventions: Drug: Single intravenous bolus of placebo at the onset of resuscitation

INTERVENTIONS:
Drug: Single intravenous bolus of cyclosporine A (2.5 mg/kg) at the onset of resuscitation — cardio-pulmonary resuscitation usual care of cardiac arrest
  Arms: Cyclosporine A
Drug: Single intravenous bolus of placebo at the onset of resuscitation — cardio-pulmonary resuscitation usual care of cardiac arrest
  Arms: Control

SUMMARY:
Cardiac arrest (CA) is a public health problem in industrialized countries. The prognosis of these patients remains poor with significant mortality and severe neurological sequelae in survivors.

The objective of the present study is to determine whether cyclosporine can improve patient clinical outcome after shockable CA. 520 patients with CA will be entered into a multicentre, randomized, placebo-controlled study. They will receive one single injection of cyclosporine (or placebo) prior to resuscitation. The incidence of the combined endpoint (mortality, irreversible brain damage informations such as bilateral abolition of N20 wave or absent motor response or extension to the nociceptive stimulation…) will be assessed 7 days after CA.

ELIGIBILITY:
Inclusion Criteria:

* Witnessed out-of-hospital cardiac arrest
* Shockable cardiac rhythm at first medical contact (ventricular fibrillation, ventricular tachycardia)

Exclusion Criteria:

* Evidence of trauma
* Evidence of pregnancy
* Duration of no flow more than 30 minutes
* Rapidly fatal underlying disease
* Allergy to cyclosporin A

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Combined incidence of all-cause mortality and irreversible brain damage status | 7 days
  the presence of irreversible brain damage is defined by the bilateral abolition of the N20 wave on somatosensory evoked potentials recordings or the absence of motor response or extension to painful stimuli on the Glasgow Coma Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Argaud, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hopital Cardiologique, Bron, France

IPD SHARING:
Plan to Share IPD: No